CLINICAL TRIAL: NCT00116116
Title: Daily Antiretroviral Therapy (DART-II): An Open-Label, Single-Arm, Prospective, Multicenter Clinical Trial To Evaluate the Efficacy and Safety fo Stavudine Extended Release (d4T XR) in Combination With Lamivudine (3TC) and Efavirenz (EFV) Once Daily in Anti-Retroviral Therapy (ART) Naive HIV-Infected Subjects
Brief Title: DART II - A Phase IV Study of 3 Antiretroviral Medicines in Combination, in HIV Patients Who Have Not Been Previously Treated With Antiretroviral Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI455-131
Record Dates: First submitted 2005-06-27; First posted 2005-06-28 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections; AIDS
Keywords: HIV/AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — efavirenz; Lamivudine

INTERVENTIONS:
Drug: efavirenz, stavudine extended release, lamivudine

SUMMARY:
The purpose of this study is to evaluate whether a therapy with an all once daily regimen of stavudine extended release (d4T XR), lamivudine (3TC), and efavirenz (EFV) leads to improved outcomes, as measured by viral load, CD4 counts, adherence, safety, and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older infected with HIV and weigh at least 40 kg.
* Plasma HIV RNA viral load of 1000 copies/mL or greater and CD4 count of 100 cells/mL or greater.
* Be willing to use two forms of contraception throughout study.
* No previous exposure to antiretroviral (ARV) drugs

Exclusion Criteria:

* Pregnancy or breastfeeding
* Physical or psychiatric disability
* Proven or suspected acute hepatitis within 30 days prior to study entry
* Active AIDS-defining opportunistic infection or disease
* History of acute or chronic pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2002-03; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Estimate efficacy of d4T-XR/3TC/EFV given QD determined by
proportion of patients with plasma HIV RNA < 400 copies/mL after 48 weeks

SECONDARY OUTCOMES:
Evaluate proportion of patients with plasma HIV RNA < 400 copies/mL at Weeks 24, 48, 72, and 96
Evaluate the proportion of patients with plasma HIV RNA < 50 copies/mL at Weeks 24, 48, 72, and 96
Determine viral suppression of plasma HIV RNA change in baseline at week 48
Determine proportion of patients whose HIV viral load doesn't drop to undetectable level within 24 weeks of therapy initiation
Evaluate time to undetectable plasma HIV RNA
Evaluate proportion of patients demonstrating virologic breakthrough
Evaluate proportion of patients demonstrating virologic failure
Evaluate time to virologic breakthrough and virologic failure
Measure magnitude and durability of changes in CD4 cell counts
Evaluate patient adherence with QD regimen using pill counts and AMAF
Determine pattern and emergence of HIV genotype resistance mutations in subjects experiencing virologic failure
Explore QoL changes using MOS-HIV health survey
Evaluate safety and tolerability of QD regimen

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Local Institution, Bakersfield, California
  - Local Institution, San Francisco, California
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Miami, Florida
  - Local Institution, New York, New York
  - Local Institution, Greenville, North Carolina
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Dallas, Texas

REFERENCES:
- [Background] Jayaweera D, Dejesus E, Nguyen KL, Grimm K, Butcher D, Seekins DW. Virologic suppression, treatment adherence, and improved quality of life on a once-daily efavirenz-based regimen in treatment-Naive HIV-1-infected patients over 96 weeks. HIV Clin Trials. 2009 Nov-Dec;10(6):375-84. doi: 10.1310/hct1006-375. PMID 20133268
- [Derived] Nunes EP, Santini de Oliveira M, Mercon M, Zajdenverg R, Faulhaber JC, Pilotto JH, Ribeiro JE, Norton M, Schechter M. Monotherapy with Lopinavir/Ritonavir as maintenance after HIV-1 viral suppression: results of a 96-week randomized, controlled, open-label, pilot trial (KalMo study). HIV Clin Trials. 2009 Nov-Dec;10(6):368-74. doi: 10.1310/hct1006-368. PMID 20133267